CLINICAL TRIAL: NCT01943396
Title: Rationalization of the Systemic Treatment of Age-related Macular Degeneration With Rheohemapheresis (RHF)
Brief Title: Treatment of AMD With Rheohemapheresis /RHF/
Acronym: TARHF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital Hradec Kralove (Other)
Responsible Party: Principal Investigator, Karel Antos, Deputy director, University Hospital Hradec Kralove
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: FNHK2013/01; IGA-NT14037-4/2013 (Other Grant/Funding Number: IGA, Ministry of Health, CZ)
Record Dates: First submitted 2013-06-20; First posted 2013-09-17 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Age Related Macular Degeneration
Keywords: age-related macular degeneration; AMD; rheohemapheresis; plasma filtration; electroretinography; ERG; multifocal ERG; double plasma filtration
MeSH Terms: conditions — Macular Degeneration | interventions — Plasmapheresis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rheohemapheresis (Experimental): Each treated patient will receive a series of 8 rheohemaphereses (cascade filtration) within 10 weeks. Best-corrected visual acuity, electroretinography and drusenoid retinal pigment epithelium detachment area will be examined. Changes of selected special immunologic parameters will be measured.
  Interventions: Procedure: rheohemapheresis
- without rheohemapheresis (No Intervention): Into the group the patients will be randomized with the same disease but without rheohemapheresis

INTERVENTIONS:
Procedure: rheohemapheresis — Each treated patient will receive a series of 8 rheohemaphereses (cascade filtration) within 10 weeks. One plasma volume will be washed.
  Other Names: rheopheresis; double plasma filtration; cascade filtration
  Arms: Rheohemapheresis

SUMMARY:
In this research rheohemapheresis will be used for the treatment of patients with high-risk dry form of age-related macular degeneration. Correction of rheologic parameters and activation of retinal functional reserves after the therapy will positively influence functional condition of retina. The newest special electrophysiologic methods will be used to determine retinal changes in time. The investigators will also evaluate some important immunologic factors and complement changes as well as define indication criteria more precisely.

DETAILED DESCRIPTION:
With optimized therapeutic protocol we would prevent progression of the dry form of AMD into its devastating wet form and stabilize the situation. We suppose that retinal morphologic and functional conditions would improve in a high percentage of patients. Also possible technical and economic savings would not be less important with our own therapeutic protocol, especially, when blindness could be prevented.

ELIGIBILITY:
Inclusion Criteria:

Patients with AMD in the stage of soft drusen, grade 1-3 according to European Eye Study (EURYEYE) (see reference No 1), body weight over 50 Kilo and with other feasible indications for aphereses therapy (peripheral veins allowing vascular access to establish the extracorporal circuit).

-

Exclusion Criteria:

* Study eye with exudative AMD
* Study eye with concomitant retinal or choroidal disorder other than AMD
* Study eye with significant central lens opacities and/or conditions that limit the view of the fundus
* uncontrolled diabetes, uncontrolled arterial hypertension
* insufficient antecubital venous access
* haemato-oncological malignancies
* patients who are unwilling to adhere to visit examination schedules . poor general condition (serious diseases - infections,cardiovascular or cerebral insufficience, severe IHD)

Max Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2013-09; Primary Completion 2016-05 (Actual); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Electroretinography | 2.5 years
  Evaluation of functional changes in single retinal layers and areas by newest special electrophysiologic methods

SECONDARY OUTCOMES:
immunologic parameters changes | 2.5 years
  To verify till undescribed changes of complement, some cytokines,factors monitoring endothelial function, and apoptosis markers, important for rapid repair of retinal revitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Milan Blaha, Prof, MD, Principal Investigator — Charles University, Medical Faculty and Faculty Hospital, 50005 Hradec Kralove, CZ
Locations (1):
- Faculty Hospital, Hradec Králové, Czechia

REFERENCES:
- [Background] Augood C, Fletcher A, Bentham G, Chakravarthy U, de Jong PT, Rahu M, Seland J, Soubrane G, Tomazzoli L, Topouzis F, Vioque J, Young I. Methods for a population-based study of the prevalence of and risk factors for age-related maculopathy and macular degeneration in elderly European populations: the EUREYE study. Ophthalmic Epidemiol. 2004 Apr;11(2):117-29. doi: 10.1076/opep.11.2.117.28160. PMID 15255027
- [Background] Blaha M, Cermanova M, Blaha V, Blazek M, Maly J, Siroky O, Solichova D, Filip S, Rehacek V. Safety and tolerability of long lasting LDL-apheresis in familial hyperlipoproteinemia. Ther Apher Dial. 2007 Feb;11(1):9-15. doi: 10.1111/j.1744-9987.2007.00450.x. PMID 17309569
- [Background] Blaha M, Zadak Z, Blaha V, Andrys C, Havel E, Vyroubal P, Blazek M, Filip S, Lanska M, Maly J. Extracorporeal LDL cholesterol elimination (25 years of experience in CZ). Atheroscler Suppl. 2009 Dec 29;10(5):17-20. doi: 10.1016/S1567-5688(09)71804-5. PMID 20129368
- [Background] Borberg H. 26 years of LDL--apheresis: a review of experience. Transfus Apher Sci. 2009 Aug;41(1):49-59. doi: 10.1016/j.transci.2009.05.013. Epub 2009 Jun 25. PMID 19559652
- [Background] Klein R, Klein BE, Knudtson MD, Meuer SM, Swift M, Gangnon RE. Fifteen-year cumulative incidence of age-related macular degeneration: the Beaver Dam Eye Study. Ophthalmology. 2007 Feb;114(2):253-62. doi: 10.1016/j.ophtha.2006.10.040. PMID 17270675
- [Background] Friedman E. The pathogenesis of age-related macular degeneration. Am J Ophthalmol. 2008 Sep;146(3):348-9. doi: 10.1016/j.ajo.2008.05.017. No abstract available. PMID 18724980
- [Background] Klingel R, Fassbender C, Fassbender T, Gohlen B. Clinical studies to implement Rheopheresis for age-related macular degeneration guided by evidence-based-medicine. Transfus Apher Sci. 2003 Aug;29(1):71-84. doi: 10.1016/S1473-0502(03)00101-0. PMID 12877897
- [Background] Klingel R, Fassbender C, Heibges A, Koch F, Nasemann J, Engelmann K, Carl T, Meinke M, Erdtracht B. RheoNet registry analysis of rheopheresis for microcirculatory disorders with a focus on age-related macular degeneration. Ther Apher Dial. 2010 Jun;14(3):276-86. doi: 10.1111/j.1744-9987.2010.00807.x. PMID 20609179
- [Background] Koss MJ, Kurz P, Tsobanelis T, Lehmacher W, Fassbender C, Klingel R, Koch FH. Prospective, randomized, controlled clinical study evaluating the efficacy of Rheopheresis for dry age-related macular degeneration. Dry AMD treatment with Rheopheresis Trial-ART. Graefes Arch Clin Exp Ophthalmol. 2009 Oct;247(10):1297-306. doi: 10.1007/s00417-009-1113-7. Epub 2009 Jul 23. PMID 19629514
- [Background] Rencová E., Bláha M., Rozsíval ry form age related macular degeneration with rheohemotherapy. (In Czech.) In Trendy soudobé oftalmologie 7. Praha: Galén, 2011, s. 16-31. ISBN 978- 80-7262- 691-5.
- [Background] Rencova E, Blaha M, Studnicka J, Blazek M, Blaha V, Dusova J, Maly J, Kyprianou G, Vasatko T, Langrova H. Haemorheopheresis could block the progression of the dry form of age-related macular degeneration with soft drusen to the neovascular form. Acta Ophthalmol. 2011 Aug;89(5):463-71. doi: 10.1111/j.1755-3768.2009.01710.x. Epub 2010 Jan 22. PMID 20102350
- [Background] Troutbeck R, Al-Qureshi S, Guymer RH. Therapeutic targeting of the complement system in age-related macular degeneration: a review. Clin Exp Ophthalmol. 2012 Jan-Feb;40(1):18-26. doi: 10.1111/j.1442-9071.2011.02581.x. PMID 22304025